CLINICAL TRIAL: NCT03835702
Title: Impact of a Novel Sleep Apnea Management Group Intervention on Positive Airway Pressure Adherence: A Randomized Controlled Trial
Brief Title: SAMPAP Trial -Impact of a Novel Sleep Apnea Management Group Intervention on Positive Airway Pressure Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: ResMed (Industry)
Responsible Party: Principal Investigator, Nancy Foldvary-Schaefer, Staff, Neurologic Institute, Sleep Disorder Center, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-110
Record Dates: First submitted 2019-01-25; First posted 2019-02-08 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-08

CONDITIONS: Sleep Apnea
Keywords: PAP; Group; PAP adherence
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care with non-sleep provider (No Intervention): Participant will continue the follow up for sleep apnea with the non-sleep provider
- SAM Clinic Intervention (Experimental): Participants will attend a sleep apnea management group based intervention to improve PAP adherence.
  Interventions: Other: SAM Clinic Intervention

INTERVENTIONS:
Other: SAM Clinic Intervention — SAM Clinic is a sleep provider led team comprised of either a sleep clinician or sleep nurse practitioner along with sleep nurses and or durable medical equipment representative. The provider interacts with each patient personally. Various modes of trouble shooting of PAP related issues are tailored to solve PAP adherence issues including mask complaints, nasal issues, pressure intolerance, anxiety, and other related barriers to PAP adherence. When the provider is seeing patients individually other patients have the opportunity to interact and offer informal interpersonal support to other participants in dealing with similar PAP issues. The provider makes an individualized follow-up plan for each patient, which may include another SAM visit or referral back to the non-sleep provider.
  Arms: SAM Clinic Intervention

SUMMARY:
This randomized controlled trial will evaluate people who have moderate-to-severe obstructive sleep apnea (OSA), and have been newly prescribed a Positive Airway Pressure (PAP) machine. Patients with suboptimal adherence, defined by the Center of Medicare and Medicaid criteria (<70 % usage and <4 hours of average daily PAP usage) will be identified. The purpose of this research is to examine the impact of the sleep apnea management (SAM) grouped based-intervention on positive airway pressure adherence and patient report outcomes questionnaires (quality of life, daytime sleepiness and depressive symptoms) and PAP barrier questionnaire compared to a patient group managed by regular non-sleep prescribing provider.

DETAILED DESCRIPTION:
The research involves collection of information from the medical record and PAP adherence collection website and completion of a survey at several time points. The survey asks questions about their experience with the therapy, quality of life, daytime sleepiness and depressive symptoms. The participants will also be provided with some literature on sleep hygiene.

Participants will be randomized to one of two groups, Sleep Apnea Management (SAM) Clinic or Usual Care with the non-sleep provider.

Questionnaires. These questionnaires are the Epworth Sleepiness Scale which measures daytime sleepiness, Patient Health Questionnaire which is a 9-item depression scale that provides psychometric measurement of depression, the PAP Barrier Questionnaire, the PROMIS Global Health, a 10-item questionnaire measuring patient reported health status for physical, mental and social well-being, The PROMIS Sleep Related Impairment, 8-item questionnaire used to identify problems in sleep the affect overall quality of sleep and the PROMIS Fatigue, another 8-item questionnaire that evaluates self-reported symptoms of tiredness that affect daily activities and functioning.

If randomized to Sleep Apnea Management (SAM) Clinic patients will be scheduled to attend the SAM Clinic. The SAM is a group clinic created to address challenges in PAP management by promoting adherence by providing access to problem-solving of PAP therapy issues. This allows patients with common problems and needs to have direct access to sleep medicine providers, sleep nurse practitioners, sleep nurses and/or durable medical equipment (DME) representatives all in one room in order to receive the most efficient service.

The questionnaires will be completed at baseline (randomization visit), after 1 month, and again at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Moderate to severe OSA (apnea hypopnea index (AHI)≥15 events/hr) on polysomnogram (PSG)
* Followed by non-sleep providers for OSA (mainly primary care providers)
* New PAP set up < 1 month
* Sub-optimal PAP adherence by objective PAP adherence data (<70 % usage and <4 hours of average PAP usage)

Exclusion Criteria:

* Central sleep apnea (>50% apneas are central) and/or presence of Cheyne-Stokes breathing
* Pregnant women
* Patients on supplemental oxygen
* Patients not able to attend SAM clinic
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Hours of PAP usage (>4 hours) in last 4 weeks and at 12 weeks. | Baseline to 3 month follow up
  To examine the impact of the sleep apnea management (SAM) group-based intervention on Positive Airway Pressure (PAP) adherence compared to a patient group managed by non-sleep medicine physicians (patients who follow usual care and are receptive to the SAM Clinic but do not participate in a SAM group) on changes from baseline to 1 and 3 months in those with moderate to severe OSA with suboptimal PAP adherence.
  Greater than 4 hours average daily use is considered adherent.
Percent days of PAP use in last 4 weeks and at 12 weeks. | Baseline to 3 month follow up
  To examine the impact of the sleep apnea management (SAM) group-based intervention on Positive Airway Pressure (PAP) adherence compared to a patient group managed by non-sleep medicine physicians (patients who follow usual care and are receptive to the SAM Clinic but do not participate in a SAM group) on changes from baseline to 1 and 3 months in those with moderate to severe OSA with suboptimal PAP adherence.
  Greater than 70% usage of days used is considered adherent.

SECONDARY OUTCOMES:
Measure changes in daytime sleepiness at 4 weeks and then at 12 weeks in PAP adherence group and in usual care group in study sample. | Baseline to 3 month follow up
  To examine and compare changes in patient reported outcomes daytime sleepiness between the SAM Clinic and the usual care arms from baseline to 1 and 3 months in those with moderate to severe OSA with suboptimal PAP adherence. To examine the correlation between changes in daytime sleepiness to changes in PAP adherence at each time point (secondary analyses).
  The Epworth Sleepiness Scale (ESS) is an 8-question scale that measures subjective daytime sleep propensity. Each question is scored on a scale of 0-3, with a total score possible of 0-24. Greater scores indicate greater daytime sleep propensity, with a score of ≥10 indicating excessive daytime sleep propensity.
  Investigators hypothesize that greater improvement in daytime sleepiness will be noted with the SAM clinic intervention compared to usual care.
Measure changes in depressive symptoms at 4 weeks and then at 12 weeks in PAP adherence group and in usual care group in study sample. | Baseline to 3 month follow up
  To compare changes in patient reported outcomes depressive symptoms between the SAM Clinic and the usual care arms from baseline to 1 and 3 months in those with moderate to severe OSA with suboptimal PAP adherence. To examine the correlation between changes in depressive symptoms to changes in PAP adherence at each time point (secondary analyses). The Patient Health Questionnaire 9 (PHQ-9) is a self-administered survey that assesses each of the 9 DSM-IV criteria for depression in a separate question. Each question is scored from 0-3, with a total possible score of 0-27. Higher scores indicate greater severity of depressive symptoms; a score of 20-27 is indicative of severe depressive symptoms warranting active treatment, 15-19 moderately severe warranting active treatment, 10-14 moderate, 5-9 mild, and 0-4 none/minimal depressive symptoms.
  Investigators hypothesize that greater improvement in depressive symptoms will be noted with the SAM clinic intervention compared to usual care.
Measure changes in global health measures at 4 weeks and then at 12 weeks in PAP adherence group and in usual care group in study sample. | Baseline to 3 month follow up
  To compare changes in patient reported outcomes global health between the SAM Clinic and the usual care arms from baseline to 1 and 3 months in those with moderate to severe OSA with suboptimal PAP adherence. To examine the correlation between changes in global health to changes in PAP adherence at each time point (secondary analyses). The PROMIS Global Health (10 questions) short form measures health. Higher score indicate greater perceived health. The raw sum score is rescaled by a t-score into a standardized score, where a standard score of 50 is the general population average (with a standard deviation of 10). If not all questions were answered, a raw score can be calculated (and later standardized) from the following formula: (Score sum of questions answered * number of questions on the form) ÷Number of questions answered.
  Investigators hypothesize that greater improvement in global health will be noted with the SAM clinic intervention compared to usual care.
Measure changes in fatigue measures at 4 weeks and then at 12 weeks in PAP adherence group and in usual care group in study sample. | Baseline to 3 month follow up
  To compare changes in patient reported outcomes in fatigue between the SAM Clinic and the usual care arms from baseline to 1 and 3 months in those with moderate to severe OSA with suboptimal PAP adherence. To examine the correlation between changes in fatigue to changes in PAP adherence at each time point (secondary analyses). The PROMIS Fatigue (8 questions) short form measures fatigue. Higher score indicate greater perceived fatigue. The raw sum score is rescaled by a t-score into a standardized score, where a standard score of 50 is the general population average (with a standard deviation of 10). If not all questions were answered, a raw score can be calculated (and later standardized) from the following formula: (Score sum of questions answered * number of questions on the form) ÷Number of questions answered.
  Investigators hypothesize that greater improvement in fatigue will be noted with the SAM clinic intervention compared to usual care.
Measure changes in sleep related impairment measures at 4 weeks and then at 12 weeks in PAP adherence group and in usual care group in study sample. | Baseline to 3 month follow up
  Compare changes in patient reported outcomes in sleep impairment between the SAM Clinic and the usual care arms from baseline to 1 and 3 months in those with moderate to severe OSA with suboptimal PAP adherence. To examine the correlation between changes in sleep impairment to changes in PAP adherence at each time point (secondary analyses). The PROMIS Sleep Related Impairment form measures sleep impairment. Higher score indicate greater perceived impairment. The raw sum score is rescaled by a t-score into a standardized score, where a standard score of 50 is the general population average (with a standard deviation of 10). If not all questions were answered, a raw score can be calculated (and later standardized) from the following formula: (Score sum of questions answered * number of questions on the form) ÷Number of questions answered.
  Investigators hypothesize that greater improvement in sleep impairment will be noted with the SAM clinic intervention compared to usual care.

OTHER OUTCOMES:
Changes in PAP Barrier questionnaire (eg. mask fit, nasal congestion, pressure intolerance) from baseline to 1 month and 3 month follow up. | Baseline to 3 month follow up
  Examine the impact of the SAM Clinic on changes in barriers to PAP adherence compared to usual care from baseline contact to 3 months in those with moderate to severe OSA with suboptimal PAP adherence.
  The Barriers questionnaire is a 12-question scale that measures subjective barriers to using a PAP machine. Each question is scored on a scale of 0-1, with a total score possible of 0-12. Greater scores indicate greater difficulty with wearing a PAP machine. Each yes answer can be addressed to improve the patient's use of the PAP.
  Investigators hypothesize that the SAM Clinic intervention will be able to address PAP barriers more effectively compared to usual care. This questionnaire is in the yes/no format. This questionnaire is in the survey that will be completed by the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Heinzinger, DO, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehra R. Sleep apnea ABCs: airway, breathing, circulation. Cleve Clin J Med. 2014 Aug;81(8):479-89. doi: 10.3949/ccjm.81gr.14002. PMID 25085986
- [Background] McEvoy RD, Antic NA, Heeley E, Luo Y, Ou Q, Zhang X, Mediano O, Chen R, Drager LF, Liu Z, Chen G, Du B, McArdle N, Mukherjee S, Tripathi M, Billot L, Li Q, Lorenzi-Filho G, Barbe F, Redline S, Wang J, Arima H, Neal B, White DP, Grunstein RR, Zhong N, Anderson CS; SAVE Investigators and Coordinators. CPAP for Prevention of Cardiovascular Events in Obstructive Sleep Apnea. N Engl J Med. 2016 Sep 8;375(10):919-31. doi: 10.1056/NEJMoa1606599. Epub 2016 Aug 28. PMID 27571048
- [Background] Weaver TE. Adherence to positive airway pressure therapy. Curr Opin Pulm Med. 2006 Nov;12(6):409-13. doi: 10.1097/01.mcp.0000245715.97256.32. PMID 17053489
- [Background] Likar LL, Panciera TM, Erickson AD, Rounds S. Group education sessions and compliance with nasal CPAP therapy. Chest. 1997 May;111(5):1273-7. doi: 10.1378/chest.111.5.1273. PMID 9149582
- [Background] Lewis KE, Bartle IE, Watkins AJ, Seale L, Ebden P. Simple interventions improve re-attendance when treating the sleep apnoea syndrome. Sleep Med. 2006 Apr;7(3):241-7. doi: 10.1016/j.sleep.2005.09.007. Epub 2006 Mar 24. PMID 16564210
- [Background] Lettieri CJ, Walter RJ. Impact of group education on continuous positive airway pressure adherence. J Clin Sleep Med. 2013 Jun 15;9(6):537-41. doi: 10.5664/jcsm.2742. PMID 23772185
- [Background] Walia HK, Griffith SD, Thompson NR, Moul DE, Foldvary-Schaefer N, Mehra R. Impact of Sleep-Disordered Breathing Treatment on Patient Reported Outcomes in a Clinic-Based Cohort of Hypertensive Patients. J Clin Sleep Med. 2016 Oct 15;12(10):1357-1364. doi: 10.5664/jcsm.6188. PMID 27568910
- [Background] Walia HK, Thompson NR, Katzan I, Foldvary-Schaefer N, Moul DE, Mehra R. Impact of Sleep-Disordered Breathing Treatment on Quality of Life Measures in a Large Clinic-Based Cohort. J Clin Sleep Med. 2017 Nov 15;13(11):1255-1263. doi: 10.5664/jcsm.6792. PMID 28992832
- [Background] Aurora RN, Collop NA, Jacobowitz O, Thomas SM, Quan SF, Aronsky AJ. Quality measures for the care of adult patients with obstructive sleep apnea. J Clin Sleep Med. 2015 Mar 15;11(3):357-83. doi: 10.5664/jcsm.4556. PMID 25700878
- [Background] Johns MW. Reliability and factor analysis of the Epworth Sleepiness Scale. Sleep. 1992 Aug;15(4):376-81. doi: 10.1093/sleep/15.4.376. PMID 1519015
- [Background] Spitzer RL, Williams JB, Kroenke K, Hornyak R, McMurray J. Validity and utility of the PRIME-MD patient health questionnaire in assessment of 3000 obstetric-gynecologic patients: the PRIME-MD Patient Health Questionnaire Obstetrics-Gynecology Study. Am J Obstet Gynecol. 2000 Sep;183(3):759-69. doi: 10.1067/mob.2000.106580. PMID 10992206
- [Background] Weaver TE, Laizner AM, Evans LK, Maislin G, Chugh DK, Lyon K, Smith PL, Schwartz AR, Redline S, Pack AI, Dinges DF. An instrument to measure functional status outcomes for disorders of excessive sleepiness. Sleep. 1997 Oct;20(10):835-43. PMID 9415942
- [Background] Bakker JP, Wang R, Weng J, Aloia MS, Toth C, Morrical MG, Gleason KJ, Rueschman M, Dorsey C, Patel SR, Ware JH, Mittleman MA, Redline S. Motivational Enhancement for Increasing Adherence to CPAP: A Randomized Controlled Trial. Chest. 2016 Aug;150(2):337-45. doi: 10.1016/j.chest.2016.03.019. Epub 2016 Mar 24. PMID 27018174
- [Background] Lachin JM. Introduction to sample size determination and power analysis for clinical trials. Control Clin Trials. 1981 Jun;2(2):93-113. doi: 10.1016/0197-2456(81)90001-5. PMID 7273794

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT03835702/Prot_SAP_000.pdf